CLINICAL TRIAL: NCT00069706
Title: Phase II Safety and Efficacy Study to Evaluate a Glaucoma Therapy in Open-angle Glaucoma or Ocular Hypertension Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-03-25
Record Dates: First submitted 2003-09-30; First posted 2003-10-06 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: open-angle; glaucoma; ocular; hypertension; POAG
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension | interventions — AL-12182; Ophthalmic Solutions; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- AL-12182 0.003% (Experimental): One drop in the study eye(s) once daily at approximately 8 a.m. for 14 days
  Interventions: Drug: AL-12182 0.003% Ophthalmic Solution
- AL-12182 Solution Vehicle (Placebo Comparator): One drop in the study eye(s) once daily at approximately 8 a.m. for 14 days
  Interventions: Other: AL-12182 Ophthalmic Solution Vehicle
- Latanoprost (Active Comparator): One drop in the study eye(s) once daily at approximately 8 a.m. for 14 days
  Interventions: Drug: Latanoprost 0.005% Ophthalmic Solution
- AL-12182 0.01% (Experimental): One drop in the study eye(s) once daily at approximately 8 a.m. for 14 days
  Interventions: Drug: AL-12182 0.01% Ophthalmic Solution
- AL-12182 0.03% (Experimental): One drop in the study eye(s) once daily at approximately 8 a.m. for 14 days
  Interventions: Drug: AL-12182 0.03% Ophthalmic Solution

INTERVENTIONS:
Drug: AL-12182 0.003% Ophthalmic Solution — Investigational ophthalmic solution intended for the treatment of open-angle glaucoma or ocular hypertension
  Arms: AL-12182 0.003%
Other: AL-12182 Ophthalmic Solution Vehicle — Placebo
  Arms: AL-12182 Solution Vehicle
Drug: Latanoprost 0.005% Ophthalmic Solution — Commercially marketed ophthalmic solution intended for the treatment of open-angle glaucoma or ocular hypertension
  Arms: Latanoprost
Drug: AL-12182 0.01% Ophthalmic Solution — Investigational ophthalmic solution intended for the treatment of open-angle glaucoma or ocular hypertension
  Arms: AL-12182 0.01%
Drug: AL-12182 0.03% Ophthalmic Solution — Investigational ophthalmic solution intended for the treatment of open-angle glaucoma or ocular hypertension
  Arms: AL-12182 0.03%

SUMMARY:
The purpose of this study is to determine the safety and IOP-lowering ability of a glaucoma therapy in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Diagnosis of open-angle glaucoma or ocular hypertension.
* LogMAR visual acuity not worse than 0.6.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Clinically relevant ophthalmic or systemic conditions.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2003-07; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure (IOP)